CLINICAL TRIAL: NCT03953001
Title: Effect of a Vibration System on Pain Reduction During Injection of Local Dental Anaesthesia in Children: a Randomized Controlled Clinical Trial
Brief Title: Effect of a Vibration System on Pain Reduction During Injection of Local Dental Anaesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Jehan AlHumaid, Associate Professor, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JH123456
Record Dates: First submitted 2019-03-29; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Local Anaesthetic; Dental Anxiety
MeSH Terms: interventions — Lidocaine; Epinephrine; Anesthetics, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Buzzy (Experimental): Buzzy was used during Maxillary anesthetic infiltration injection with 2%lidocaine with 1:50,000 epinephrine after topical application with 20% Benzocaine topical gel.
  Interventions: Device: Adminstration Technique using Buzzy external distractor; Drug: 2% Lidocaine with 1:50,000 epinephrine; Drug: Topical Anesthetic
- Control (Active Comparator): Maxillary anesthetic infiltration injection with 2%lidocaine with 1:50,000 epinephrine after topical application with 20% Benzocaine topical gel only.
  Interventions: Drug: 2% Lidocaine with 1:50,000 epinephrine; Drug: Topical Anesthetic

INTERVENTIONS:
Device: Adminstration Technique using Buzzy external distractor — External application of Buzzy distractor during administration of dental anesthetic
  Arms: Buzzy
Drug: 2% Lidocaine with 1:50,000 epinephrine — Local Dental anesthetic infiltration
Drug: Topical Anesthetic — 20% Benzocaine gel was applied on the area of infiltration

SUMMARY:
The study assesses the effect of a new vibration system on pain reduction during the injection of local anesthesia. Children undergoing dental treatment are allocated to two groups; one receiving the Buzz, a vibration system and another group receiving nothing. Pain during injection of local anesthetic is assessed using a validated tool in addition to assessment of child cooperation during treatment.

DETAILED DESCRIPTION:
Eligibility of children for inclusion into the study will be assessed followed by random sequence generation and randomization into one of the two study group and allocation concealment. Topical anaesthesia will be administered to the two groups followed by implementation of the vibration system in the test group. . Behavior and pain will assessed at the time of injection.

ELIGIBILITY:
Inclusion Criteria:

1. Children 5-12 years of age.
2. Positive or definitely positive behavior on Frankl scale.6
3. Children receiving treatment on the dental chair.
4. Free from allergies to topical anesthetic used in the study.
5. Parental consent for child participation in the study.

Exclusion Criteria:

1. Those in need of treatment under general anesthesia will be excluded from the study.
2. Children with allergies from topical anesthesia

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Self Reported pain intensity: Visual analogue scale (VAS) of pain intensity | Procedure (immediately after the administration of Dental anesthesia)
  Self reported pain intensity before the injection and directly after the injection. Each child scored pain intensity twice, one before the injection and one directly after the injection (0=no pain; 10=Very painful).

SECONDARY OUTCOMES:
Parents Perception for the child tolerance of pain; Observational Pain rating scale | Procedure (immediately after the administration of Dental anesthesia.)
  The parents were asked about the reaction and attitude of the child during the dental anesthesia administration. Parents rated the child ability to tolerate pain with (0=Didn't Tolerate and 10= Tolerated with a smile)
External observation for Facial and Physical expression. Using Sounds, Eyes, and Motor (SEM) scale (RANGE 0-9). | Procedure (immediately during and after the administration of Dental anesthesia.)
  Video was recorded for each child before, during and after the administration of local anesthesia. Each video was assessed by an external calibrated evaluator to score each child response. SEM (0=Comfortable, with no sound, no eye signs of discomfort and Hands are relaxed, no apparent body tenseness, 9= Painful, with verbal complain, crying tears and moving the hands to make aggressive physical contact and pulling the head away. The lowest record mean the child was comfortable and the higher the score mean the child experienced discomfort.
Faces Legs Activity Cry Consolability (FLACC) Scale (RANGE 0-10) | Procedure (immediately during and after the administration of Dental anesthesia.)
  Video was recorded for each child before, during and after the administration of local anesthesia. Each video was assessed by an external calibrated evaluator to score each child response. FLACC (0=The child did not express any facial discomfort with normal legs position no abnormal activity, not crying and relaxed. The highest score 10= Child experienced discomfort, moving his legs jerking crying and difficult to console. The lowest record mean the child was comfortable and the higher the score mean the child experienced discomfort.

CONTACTS AND LOCATIONS:
Overall Officials: Jehan A AlHumaid, DSc, Principal Investigator — imam Abdulrahman Bin Faisal
Locations (1):
- imam adbulrahman Bin Faisal University- College of Dentistry, Dammam, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] AlHareky M, AlHumaid J, Bedi S, El Tantawi M, AlGahtani M, AlYousef Y. Effect of a Vibration System on Pain Reduction during Injection of Dental Anesthesia in Children: A Randomized Clinical Trial. Int J Dent. 2021 Jan 30;2021:8896408. doi: 10.1155/2021/8896408. eCollection 2021. PMID 33564311